CLINICAL TRIAL: NCT04345107
Title: A Phase Ib Placebo-controlled Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SY-009 After Multiple Ascending Doses in Patients With Type 2 Diabetes Mellitus
Brief Title: Multiple Ascending Doses of SY-009 in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SY009002
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- SY-009-1mg/d-1 (Experimental): 0.5mg BID. The subjects were given the drug for the first time before breakfast in D1, and then continued to take the drug daily until dinner in D7, and left after PD sample collection and safety assessment before breakfast in D8. Start at the same time as the SY-009-1mg/d-2 group. At the end of the two groups, the researchers will decide whether to move on to the next stage，2mg/d.
  Interventions: Drug: SY-009
- SY-009-1mg/d-2 (Experimental): 1mg QD.The subjects were given the drug for the first time before breakfast in D1, and then continued to take the drug daily until dinner in D7, and left after PD sample collection and safety assessment before breakfast in D8.Start at the same time as the SY-009-1mg/d-1 group. At the end of the two groups, the researchers will decide whether to move on to the next stage，2mg/d.
  Interventions: Drug: SY-009
- SY-009-2mg/d-1 (Experimental): 1mg BID.The subjects were given the drug for the first time before breakfast in D1, and then continued to take the drug daily until dinner in D7, and left after PD sample collection and safety assessment before breakfast in D8. Start at the same time as the SY-009-2mg/d-2 group. At the end of the two groups, the researchers will decide whether to move on to the next stage，4mg/d.
  Interventions: Drug: SY-009
- SY-009-2mg/d-2 (Experimental): 2mg QD.The subjects were given the drug for the first time before breakfast in D1, and then continued to take the drug daily until dinner in D7, and left after PD sample collection and safety assessment before breakfast in D8. Start at the same time as the SY-009-2mg/d-1 group. At the end of the two groups, the researchers will decide whether to move on to the next stage，4mg/d.
  Interventions: Drug: SY-009
- SY-009-4mg/d (Experimental): 2mg BID.The subjects were given the drug for the first time before breakfast in D1, and then continued to take the drug daily until dinner in D7, and left after PD sample collection and safety assessment before breakfast in D8. If the test and safety assessment of 4mg daily dose group (2mg bid) are completed and the dose termination standard is not met, the test will be terminated; if the safety assessment during or after the test reaches the dose termination standard, the study of 3mg daily dose group (1.5mg bid) will be carried out, and then the test will be terminated.
  Interventions: Drug: SY-009
- SY-009-3mg/d (Experimental): 1.5mg BID.The subjects were given the drug for the first time before breakfast in D1, and then continued to take the drug daily until dinner in D7, and left after PD sample collection and safety assessment before breakfast in D8, and then the test will be terminated.
  Interventions: Drug: SY-009
- SY-009 matching placebo (Placebo Comparator): Oral administration of the same number of tablets in the corresponding test group.
  Interventions: Drug: SY-009 matching placebo

INTERVENTIONS:
Drug: SY-009 — The subjects were admitted to the clinical trial center two days before the administration period (D-2), fasted for 10 hours overnight on the day before the Administration (D-1), and banned water for 1 hour before the administration. Take sy-009 test drug or placebo immediately before meal (QD is before breakfast, bid is before breakfast and dinner) in the morning of the first day of administration, and deliver it with not more than 200ml warm boiled water. From the day 2 (D2) to the day 7 (D7) before dinner, the oral cavity of the subjects was checked for residual drugs after each administration.
  Arms: SY-009-1mg/d-1; SY-009-1mg/d-2; SY-009-2mg/d-1; SY-009-2mg/d-2; SY-009-3mg/d; SY-009-4mg/d
Drug: SY-009 matching placebo — SY-009 matching placebo
  Arms: SY-009 matching placebo

SUMMARY:
This is a phase Ib placebo-controlled study to assess safety, tolerability, pharmacokinetics and pharmacodynamics of SY-009 after Multiple Ascending Doses in patients with Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, dose-increasing, multiple oral administration clinical trial. The planned dose escalation levels were 1, 2, 3 and 4 mg daily (6 dose groups).

After the completion of the test and safety evaluation of the initial dose of 1mg daily dose in two groups (0.5mg bid and 1mg QD), the main researchers of the team leader and the sponsor jointly determine whether to enter the 2mg daily dose study.

After the completion of the test and safety evaluation of two groups (1mg bid and 2mg QD) of 2mg daily dose, the main researchers of the group leader and the sponsor jointly determine whether to enter the 4mg daily dose study.

If the test and safety assessment of 4mg daily dose group (2mg bid) are completed and the dose termination standard is not met, the test will be terminated; if the safety assessment during or after the test reaches the dose termination standard, the study of 3mg daily dose group (1.5mg bid) will be carried out, and then the test will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* body weight of male ≥ 50kg, female ≥ 45kg, and body mass index (BMI) between 18.0 and 35.0 kg / m2 (including the threshold value) at screening;
* Have T2DM prior to entering the trial based on the disease diagnostic criteria (WHO, 1999), and currently being treated with diet and exercise only for at last 12 weeks , or no systemic treatment of diabetes (the cumulative use of antidiabetic drugs in the past 3 months has lasted no more than 2 weeks and no antidiabetic drugs has been used in the past month);
* 7% ≤ HbA1c ≤ 9.5% at screening;
* 7 mmol/L≤FPG ≤ 13.3 mmol/L at baseline;
* During the study period and within 60 days after the end of the study, the subjects has no fertility or sperm / egg donation plan and will voluntarily take effective physical contraceptive measures;
* Have given written informed consent to participate in this study, are well motivated, capable, and willing to communicate with the investigator and complete all the requirements according to the protocol.

Exclusion Criteria:

* Those who are known to be allergic to the test drug (including the auxiliary materials of the test drug) or its analogues, or who are allergic to two or more drugs, food and pollen, or who have taken SGLT1 or SGLT2 inhibitors in the past year;
* It was diagnosed as type 1 diabetes, or gestational diabetes, or other special type diabetes;
* There is enough evidence to show that there is proliferative retinopathy of active diabetes;
* History of severe hypoglycemia (such as consciousness disorder and coma caused by hypoglycemia), or history of severe unconsciousness hypoglycemia;
* Organ transplantation history, or other acquired, congenital immune system diseases, or peripheral vascular diseases with clinical significance;
* Have significant hyperglycemia symptoms, such as polyuria, polydipsia, accidental weight loss or dehydration;
* Habitual diarrhea, irritable bowel syndrome, clinically significant abnormal gastric emptying (such as gastric outlet obstruction), severe chronic gastrointestinal diseases (such as active ulcer within 6 months), long-term medication with direct impact on gastrointestinal peristalsis, or gastrointestinal surgery;
* Have obvious blood system diseases (such as aplastic anemia, myelodysplastic syndrome), or any disease causing hemolysis or red blood cell instability (such as malaria), or accompanied by hemoglobin diseases (such as sickle type red blood cell disease) that may affect the determination of HbA1c level;
* Obvious autonomic neuropathy, such as urinary retention, orthostatic hypotension, diabetic diarrhea or gastroparesis.
* History of heart failure (NYHA class Ⅲ and Ⅳ, Appendix 2), or history of acute myocardial infarction or unstable angina within 6 months before screening, or history of coronary angioplasty, coronary stent implantation or coronary bypass surgery within 6 months before screening, or recent cardiac surgery plan;
* Serious trauma, infection or operation that may affect blood glucose control occurred within one month before screening;
* In the first two months of the screening, the drug with weight control effect was used or the operation that can lead to weight instability was performed, or the drug is currently in the weight-loss plan and is not in the maintenance stage;
* Completed or withdrawn an intervention clinical trial within 3 months before screening, or is currently conducting the intervention clinical trial, or participated in other medical research activities, which is not suitable for the study according to the judgment of the researcher;
* Those who frequently drink alcohol (more than 21 units (male) and 14 units / week (female) (1 unit = 360ml beer; or 150ml wine; or 45ml white wine) in the three months before screening, or who can't stop drinking during the test;
* Those who are addicted to smoking (more than 10 cigarettes per day or the same amount of tobacco) within 3 months before screening or who cannot quit smoking (stop nicotine intake) during the trial;
* Those who lost / donated more than 400 ml blood within 3 months before screening (except female physiological blood loss), received blood transfusion or used blood products, or planned to donate blood within 1 month (30 days) after the end of the trial or during the trial;
* To screen the patients with unstable thyroid function (such as thiourea and thyroid hormone drugs) in the first 6 months, with poor control of hypothyroidism or history of hypothyroidism;
* In the first 6 months of screening, there was a history of diabetic acute metabolic complications (diabetic ketoacidosis, hyperosmotic nonketotic coma, diabetic lactate acidosis);
* In the screening period, when no pacemaker was installed, 12 lead ECG showed second degree or third degree atrioventricular block or qtcb interval prolonged more than 500 ms;
* The results of clinical laboratory examination in screening period meet any of the following criteria:

  1. Hemoglobin (Hgb) < lower limit of normal value (LLN);
  2. Aspartate transaminase (AST) or alanine transaminase (ALT) > 2 times of upper limit of normal value (ULN);
  3. Total bilirubin (TBIL) > 1.5 times the upper limit of normal value (except for known Gilbert syndrome which meets the following requirements, that is, part of bilirubin indicates that the combined bilirubin is less than 35% of total bilirubin);
  4. Triglyceride (TG) ≥ 5.7mmol/l;
  5. Estimated glomerular filtration rate < 60 ml / min (estimated by Cockroft Gault formula);
  6. Fasting C peptide < 1.0 ng / ml (333 pmol / L);
  7. Hepatitis B surface antigen, hepatitis C virus antibody, Treponema pallidum antibody or human immunodeficiency virus antibody were screened positive;
* Poor blood pressure control (SBP ≥ 160mmhg and / or DBP ≥ 100mmhg);
* Patients with history of needle syncope, blood syncope or intolerant of venipuncture;
* Those with a history of drug abuse or positive drug abuse screening;
* Patients with obvious mental disorders, epilepsy and other persons without behavioral or cognitive abilities;
* Female subjects in pregnancy, lactation, or with pregnancy intention, or positive pregnancy test (hCG test); and female subjects of childbearing age who can not take effective contraceptive measures (effective contraceptive measures include abstinence, sterilization, intrauterine device, or diaphragm method stipulated by local laws) during the test period;
* The subject may not complete the study for other reasons or the researcher thinks it should not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Maximum postprandial (breakfast, lunch, dinner) blood glucose added value | 7 days
  Compared with placebo, the maximum change in glucose from baseline at D7.
Blood glucose AUC (AUC 0-4,AUC 4-10, AUC 10-14, AUC 0-24) in different periods. | 7 days
  Compared with placebo, the mean change in glucose AUC from baseline at D7.
The Safety and tolerance of SY-009，Collecting Number of subjects with adverse events as assessed by CTCAE V5.0 | 7 days
  Number of subjects with adverse events, major adverse events, serious adverse events, abnormal Laboratory Values, abnormal vital signs, Abnormal physical examination, Abnormal ECG data，Gastrointestinal adverse reactions (diarrhea, etc.) and hypoglycemia events
C-peptide concentration changes before and after meal. | 7 days
  Compared with placebo, the mean change from baseline at D7.
The changes of insulin concentration before and after meal. | 7 days
  Compared with placebo, the mean change from baseline at D7.
GLP-1 concentration changes before and after meal. | 7 days
  Compared with placebo, the mean change from baseline at D7.
GIP concentration changes before and after meal. | 7 days
  Compared with placebo, the mean change from baseline at D7.

SECONDARY OUTCOMES:
Peak concentration (Cmax) | 1 day
  after the first dose
Peak time (Tmax) | 1 day
  after the first dose
Terminal elimination rate constant (λ z) | 1 day
  after the first dose
Terminal elimination half-life (T1 / 2) | 1 day
  after the first dose
Area under the drug time curve from 0 to the last detectable time (auc0-t) | 1 day
  after the first dose
Area under the drug time curve (auc0 - ∞) from 0 to infinite time | 1 day
  after the first dose
Auc0 - ∞ extrapolation percentage (% aucex) | 1 day
  after the first dose
Apparent clearance (CL / F) | 1 day
  after the first dose
Apparent distribution volume (VZ / F). | 1 day
  after the first dose
Steady state peak concentration (Cmax, SS). | 7 days
  After reaching steady state
Steady state peak time (Tmax, SS). | 7 days
  After reaching steady state
Steady state terminal elimination half-life (T1 / 2, SS). | 7 days
  After reaching steady state
Area under drug time curve (auc0-t, SS) from steady state 0 to last detectable time. | 7 days
  After reaching steady state
The area under the drug time curve (auc0 - ∞, SS) of steady state from 0 to infinite time. | 7 days
  After reaching steady state
Auc0 - ∞ extrapolation percentage (% aucex) | 7 days
  After reaching steady state
Accumulation ratio (rauc, rcmax) | 7 days
  After reaching steady state
Stable Valley concentration (ctrough, SS). | 7 days
  After reaching steady state

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yuncheng Central Hospital, Yuncheng, Shanxi

REFERENCES:
- [Derived] Yang H, Zhang Y, Hong Y, Wei Y, Zhu Y, Huang L, Yang Y, Sun R, Li J. Effect of SY009, a novel SGLT1 inhibitor, on the plasma metabolome and bile acids in patients with type 2 diabetes mellitus. Front Endocrinol (Lausanne). 2025 Jan 28;16:1487058. doi: 10.3389/fendo.2025.1487058. eCollection 2025. PMID 39936104
- [Derived] Huang L, Cao B, Geng Y, Zhou X, Yang Y, Ma T, Lin H, Huang Z, Zhuo L, Li J. A randomized double-blind phase Ib clinical trial of SY-009 in patients with type 2 diabetes mellitus. Eur J Pharm Sci. 2024 Jan 1;192:106644. doi: 10.1016/j.ejps.2023.106644. Epub 2023 Nov 20. PMID 37981049